CLINICAL TRIAL: NCT05246735
Title: Frequency Domain Optical Imaging of Breast Cancer
Brief Title: Frequency Domain Optical Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Keith D. Paulsen, Professor of Engineering, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00011487
Record Dates: First submitted 2022-02-16; First posted 2022-02-18 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a clinical study to evaluate MR-guided near infrared absorption and fluorescence imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided NIR (Other): Women with breast abnormalities will undergo an "optical exam" (NIR) in combination with MRI where the NIR light imaging system illuminates the breast from multiple positions covering the area of interest.
  A total of 60 women will be evaluated: 20 with breast abnormalities receiving gadolinium (Gd) contrast enhancement, 20 with breast abnormalities receiving both Gd-contrast enhancement and indocyanine green (ICG) contrast enhancement, and 20 healthy volunteers not receiving any contrast agents.
  Interventions: Diagnostic Test: MR-guided Near Infrared optical tomography

INTERVENTIONS:
Diagnostic Test: MR-guided Near Infrared optical tomography

SUMMARY:
This purpose of this clinical study to develop and test technology associated with near infrared (NIR) optical tomography of the breast (the use of light at NIR wavelengths to image the breast) as an adjunct to mammography and breast MRI.

DETAILED DESCRIPTION:
The purpose of this clinical study is to demonstrate the feasibility of NIR absorption and fluorescence imaging of the female breast when the method is guided by breast MRI. The hypotheses to be tested are:

1. MR-guided NIR absorption and fluorescence imaging of the breast is feasible in the setting of a clinical breast exam
2. MR-guided NIR absorption and fluorescence imaging of the breast provides spatial localization and contrast of a breast abnormality that is superior to NIR absorption and fluorescence tomography alone.

ELIGIBILITY:
HEALTHY VOLUNTEERS

Inclusion Criteria:

1. Female, ≥20 years old
2. Breast size and epithelial integrity adequate to allow NIR imaging exams.
3. Ability to provide written informed consent
4. No serious associated psychiatric illnesses.

Exclusion Criteria:

1. Absolute or relative contraindication to MRI:

   1. the presence of an electronic implant, such as a pacemaker
   2. the presence of a metal implant, such as an aneurysm clip
   3. claustrophobia
   4. the presence of other contraindication(s), as determined by the MRI technologists and radiologists.
2. Pregnancy

WOMEN WITH BREAST ABNORMALITIES

Inclusion:

1. Female, ≥ 20 years old.
2. Breast size and epithelial integrity adequate to allow NIR imaging exams.
3. Ability to provide written informed consent.
4. No serious associated psychiatric illnesses.
5. A recent screening mammogram that questions the presence of an abnormality, thus requiring further mammographic examination.

Exclusion:

1. Absolute or relative contraindication to MRI:

   1. the presence of an electronic implant, such as a pacemaker
   2. the presence of a metal implant, such as an aneurysm clip
   3. claustrophobia
   4. the presence of other contraindication(s), as determined by the MRI technologists and radiologists.
2. Pregnancy
3. A history of allergy to iodides
4. A GFR < 30 ml/min as determined by blood test on the day of NIR/MR imaging, or from lab results within 3 months of NIR/MR imaging.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02-01 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Compare spatial localization and contrast images of breast abnormalities from MR-guided NIR absorption and fluorescence tomography to NIR absorption and fluorescence tomography alone | During imaging and evaluation by a radiologist or medical technologist, up to 90 minute
  Women will participate in MR-guided NIR exams which include both MR and optical contrast agents. These imaging outcomes will be compared to exams where only the MR contrast agent is used as well as to exams where no contrast agents are administered.

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Paulsen, PhD, Principal Investigator — Dartmouth College

IPD SHARING:
Plan to Share IPD: No